CLINICAL TRIAL: NCT04887779
Title: Pathologist Led Intervention To Improve Psychological Outcomes and Adherence in Lung Transplant Patients
Brief Title: Pathologist Lung Transplant Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: personale shortage
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Blake Gibson, Psychiatry Resident at UPMC Western Psychiatric Hospital, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19060024
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Adherence, Patient; Psychological; Coping Skills
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Prospective, no blinding or randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patient viewing ex-planted organ and microscopy with pathologist
  Interventions: Behavioral: Pathologist intervention

INTERVENTIONS:
Behavioral: Pathologist intervention — viewing explanted organ and microscopy

SUMMARY:
Using a prospective qualitative approach, explore whether pathologist intervention is feasible as part of multimodal multidisciplinary care model for transplant patients in effecting psychological dimensions such as experience, satisfaction, or patient's understanding of their disease. Additionally, to examine if this intervention improves medication adherence.

DETAILED DESCRIPTION:
Specific Aims 1. Create post-transplant pathologist-led intervention Objective 1a: Recruit 10 patients who have undergone lung transplantation primarily for chronic obstructive pulmonary disease (COPD). Use pathologist to show gross/microscopic explanted organs.

Specific Aim 2. Assess the efficacy of intervention pilot Objective 2a: Immediate (within 1 day after pathologist intervention) phone interview to access patient's reaction, feelings, and experience with intervention and understanding of disease.

Objective 2b: 1 month later, phone interview asking questions related to medication adherence, patient experience with intervention and lung transplant overall, and patient understanding of disease. Results will be compared to first interview.

Objective 2c: Analyze Client Satisfaction Questionnaire (CSQ-8) for quality of life, Basel assessment of adherence to immunosuppressive medications scale (BAASIS) as a self report adherence measure, and conduct a mixed methods/grounded theory analysis of qualitative data (patient experience, disease understanding). This analysis will systematically identify themes, and assign these descriptive words.

Specific Aim 3: Finalize intervention protocol based on pilot testing. Objective 3a. Adjust and refine the content and process of intervention protocol based on findings of pilot study Objective 3b. Final changes will assure readiness for large scale study.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant patient, transplanted after IRB approval of study -Transplanted primarily for COPD
* English speaking
* within three months of initial transplant (prior to initial discharge)
* > 18 years old

Exclusion Criteria:

* Transplant indication other than COPD
* <18 year old
* Non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Basel Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS©) | one day after intervention and assessment for change one month later
  The Basel Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS©) was developed to assess adherence to immunosuppressive drugs in adult and adolescent transplant recipients. Initiation starts when a patient takes his/her first dose of medication. This is a binary event (yes/no). Implementation of the dosing regimen refers to "the extent to which a patient's actual dosing corresponds to the prescribed dosing regimen, from initiation until the last dose is taken" and implies a dosing history.
  Discontinuation refers to "the moment that the patient discontinues his/her medication regimen" and is assessed as a time to event. Persistence is thus the duration between time of initiation and the moment the last dose is taken. Any yes response demonstrates issues with medication adherence.
Client Satisfaction Questionnaire (CSQ-8) | one day after intervention and assessment for change one month later
  The Client Satisfaction Questionnaire is an 8 item measure of client satisfaction. An "overall score" is calculated by summing the respondent's rating (item rating) score for each scale item. Scores therefore range from 8 to 32, with higher values indicating higher satisfaction. with services with both a parent intervention versus averages of lung transplant patients.

SECONDARY OUTCOMES:
Patient understanding | one day after intervention and assessment for change one month later
  Assess if patient has gained more understanding of their condition. No specific scale used, assessed by interview.
Patient experience | one day after intervention and assessment for change one month later
  Discussing patient's overall experience. No specific scale used, assessed by interview.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Gibson, MD, Principal Investigator — University of Pittsburgh Medical Center Western Psychiatric Hospital
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No